CLINICAL TRIAL: NCT01040156
Title: Safety, Feasibility and Efficacy of Caspofungin Versus Liposomal Amphotericin B as Antifungal Prophylaxis Following Allogeneic Hematopoietic Stem Cell Transplantation in Pediatric Patients - a Retrospective Phase I/II Study
Brief Title: Antimycotic Prophylaxis in Pediatric Patients Following Allogeneic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: University Children's Hospital Tuebingen (Other)
Other Study IDs: UCHT-1209
Record Dates: First submitted 2009-12-28; First posted 2009-12-29 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Systemic Aspergillosis; Systemic Candidiasis
MeSH Terms: conditions — Systemic candidiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- LAmb
- Cas

SUMMARY:
Pediatric patients are at high risk to acquire mycotic infections following allogeneic bone marrow transplantation. In the present retrospective analysis we assess the safety and efficacy of different regimens in antimycotic prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients under the age of 18 years
* Pediatric patients after HSCT treated with caspofungin
* Pediatric patients after HSCT treated with liposomal amphotericin

Exclusion Criteria:

* Pediatric patients with uncontrolled hematological malignancies
* Pediatric patients with IFI at start of HSCT

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric patients undergoing allogeneic stem cell transplantation
Sampling Method: Non-Probability Sample
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Mueller, M.D., Principal Investigator — UCHT
Locations (1):
- University Children's Hospital, Tübingen, Germany